CLINICAL TRIAL: NCT02782117
Title: Luminopia One Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luminopia (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-AM-1C AND C-AM-1D
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: A single-arm, multi-center, open-label pilot study conducted in two phases. Phase 1 enrolled 10 participants at 1 site and phase 2 enrolled 74 participants at 9 sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Regimen A (Experimental): Treatment Regimen A will use the Luminopia device for an hour per day for 12 weeks.
  Interventions: Device: Luminopia One

INTERVENTIONS:
Device: Luminopia One — Luminopia One is a digital therapeutic that allows patients to watch videos with therapeutic modifications applied.

SUMMARY:
A single-arm, multi-center, open-label pilot study to evaluate the feasibility, safety, and efficacy of the Luminopia One digital therapeutic in improving visual acuity in a pediatric amblyopia population.

ELIGIBILITY:
Major Eligibility Criteria:

* Age 4 to <8 years (phase 1) or age 4 to <13 years (phase 2)
* Monocular amblyopia associated with anisometropia, strabismus or both combined
* Amblyopic eye best-corrected visual acuity (BCVA) 20/40 to 20/200 inclusive (0.3-1.0 logMAR)
* Fellow eye BCVA 20/25 or better (phase 1) or 20/32 or better (phase 2)
* Interocular BCVA difference ≥3 lines (≥0.3 logMAR)
* Visual acuity stability in current refractive correction (phase 2)
* Corrected distance heterotropia ≤5 prism diopters on simultaneous prism and cover test (SPCT)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Amblyopic eye best-corrected visual acuity | 12 weeks
  Electronic ATS-HOTV protocol for participants < 7 years of age and electronic ETDRS protocol for participants ≥ 7 years of age

SECONDARY OUTCOMES:
Amblyopic eye best-corrected visual acuity | 8 weeks
  Electronic ATS-HOTV protocol for participants < 7 years of age and electronic ETDRS protocol for participants ≥ 7 years of age
Amblyopic eye best-corrected visual acuity | 4 weeks
  Electronic ATS-HOTV protocol for participants < 7 years of age and electronic ETDRS protocol for participants ≥ 7 years of age
Adherence | 12 weeks
  Duration spent using the device divided by duration of treatment prescribed (objectively monitored)

CONTACTS AND LOCATIONS:
Overall Officials: David Hunter, MD PhD, Study Director — Boston Children's Hospital
Locations (9):
- United States (9):
  - Eye Physicians of Central Florida, Maitland, Florida
  - Wheaton Eye Clinic, Chicago, Illinois
  - Indiana University, Bloomington, Indiana
  - Kids Eye Care of Maryland, Frederick, Maryland
  - Children's Eye Care of Michigan, Dearborn, Michigan
  - Concord Eye Center, Concord, New Hampshire
  - Conestoga Eye, Lancaster, Pennsylvania
  - Houston Eye Associates, Houston, Texas
  - Virginia Pediatric Eye Center, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No